CLINICAL TRIAL: NCT01232881
Title: Predicting Response and Toxicity in Patients Receiving Lonafarnib for Breast Cancer: A Multicenter Genomic, Proteomic and Pharmacogenomic Correlative Study
Brief Title: Predicting Response and Toxicity in Patients Receiving Lonafarnib for Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: funding terminated
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Indiana University School of Medicine (Other); Emory University (Other)
Responsible Party: George Sledge, M.D., Hoosier Oncology Group
Other Study IDs: HOG COE-03
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumor sample submission can consist of a fresh frozen tissue sample or a formalin-fixed paraffin embedded tissue block.
  Serum is to be collected prior to the initiation of lonafarnib treatment and 28 days after the last dose of lonafarnib.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Tumor and Serum Collection: Tumor sample submission can consist of a fresh frozen tissue sample or a formalin-fixed paraffin embedded tissue block.
  Serum is to be collected prior to the initiation of lonafarnib treatment and 28 days after the last dose of lonafarnib.
  Interventions: Procedure: Tumor Sample; Procedure: Serum Sample

INTERVENTIONS:
Procedure: Tumor Sample — Tumor sample submission can consist of a fresh frozen tissue sample or a formalin-fixed paraffin embedded tissue block.
Procedure: Serum Sample — Serum is to be collected prior to the initiation of lonafarnib treatment and 28 days after the last dose of lonafarnib.

SUMMARY:
This is a tumor and serum collection study for patients with advanced breast cancer receiving treatment with lonafarnib.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Sample Collection:

* Tumor sample
* Serum sample

Treatment Regimen:

* All registered patients must be planning treatment with lonafarnib

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age > 18 years.
* Planned treatment with lonafarnib for metastatic breast cancer.
* Must consent to have a biopsy performed to obtain fresh tissue or be able to identify a formalin fixed paraffin embedded (FFPE) tissue block in which tumor samples can be obtained to complete the testing for this study.

Exclusion Criteria:

* Planned treatment with any other treatment regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be limited to patients with advanced breast cancer receiving treatment with lonafarnib.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To correlate tumor gene expression (genomic profile) with response to lonafarnib in patients with advanced breast cancer | 24 months

SECONDARY OUTCOMES:
To correlate serum and tumor proteomic profiles with response to lonafarnib | 24 months
To compare serum and tissue proteomic analyses | 24 months
To compare genomic and proteomic profiles | 24 months
To correlate toxicity and /or response with drug-specific pharmacogenomic parameters | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: George Sledge, M.D., Study Chair — Hoosier Cancer Research Network
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States

REFERENCES:
- See also: Hoosier Oncology Group Homepage — http://www.hoosieroncologygroup.org